CLINICAL TRIAL: NCT05170087
Title: Radiomic Analysis of CT and MRI Scans for Predicting Treatment Response and Clinical Outcomes in Patients With Breast, Brain, Head-neck and Gynecological Malignancies
Brief Title: Radiomic Analysis for Predicting Treatment Response and Clinical Outcomes in Malignancies
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Gregory Czarnota, Radiation Oncologist and Clinical Scientist, Sunnybrook Health Sciences Centre
Other Study IDs: 034-2020
Record Dates: First submitted 2021-11-23; First posted 2021-12-27 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer; Head and Neck Cancer; Brain Cancer; Gynecologic Cancer
MeSH Terms: conditions — Breast Neoplasms; Head and Neck Neoplasms; Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Breast malignancies: Those diagnosed with breast malignancies
- Head and Neck malignancies: Those diagnosed with head and neck malignancies
- Brain malignancies: Those diagnosed with brain malignancies
- Gynecological malignancies: Those diagnosed with gynecological malignancies

SUMMARY:
In this study, the investigators aim to undertake a retrospective analysis of CT and MRI scans for patients undergoing radiation treatment to develop radiomic signatures to predict treatment response and clinical outcomes.

DETAILED DESCRIPTION:
Imaging in oncology has widespread application with modalities like ultrasound, computed tomography (CT), magnetic resonance imaging (MRI), positron emission tomography (PET) having a well-established role particularly in diagnosis, staging, assessment of treatment response, and surveillance. With the applications of radiomics in oncology, the potential of imaging as a non-invasive biomarker in treatment response, as well as genotypic characterization, has been recognized. Radiomics has the potential to tailor way towards precision oncology with the development of biomarkers that can guide personalized treatments. In this study, the investigators aim at developing CT and MRI radiomic signatures as potential biomarkers to predict treatment response and clinical outcomes for patients treated with radiation having breast, brain, head and neck, and gynecological malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Breast, head and neck, brain, and gynecological malignancies
* Treated with radiation at Odette Cancer Centre between 2010 and 2019

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Those treated with radiation at Odette Cancer Centre between 2010 and 2019 after being diagnosed with a breast, brain, head and neck, or gynecological malignancy.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2020-03-02 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Development of imaging biomarkers in predicting treatment response for breast, brain, head-neck, and gynecological malignancies | 1 year
  Development of imaging biomarkers in predicting treatment response
Development of imaging biomarkers in predicting clinical outcomes (survival/toxicity) for breast, brain, head-neck, and gynecological malignancies | 1 year
  Development of imaging biomarkers in predicting clinical outcomes (survival/toxicity)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Czarnota, Ph.D. M.D., Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada